CLINICAL TRIAL: NCT02465021
Title: Innovation of Breakfast Cereals and Snacks for Control of Appetite and Post-Prandial Glycemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: General Mills (Industry)
Responsible Party: Principal Investigator, G. Harvey Anderson, Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 30422
Record Dates: First submitted 2015-06-03; First posted 2015-06-08 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Obesity; Diabetes
Keywords: Satiety; Food intake; Breakfast cereals/snacks; Postprandial glycemia
MeSH Terms: conditions — Obesity; Diabetes Mellitus | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Snack bar 1 (Experimental): Dietary intervention: 190 Kcal, 12g fat, 14g carbohydrate, 5g fibre, 6g sugar, 10g protein
  Interventions: Other: Dietary intervention
- Snack bar 2 (Experimental): Dietary intervention: 200 Kcal, 15g fat, 12g carbohydrate, 5g fibre, 4g sugar, 8g protein
  Interventions: Other: Dietary intervention
- Snack bar 3 (Experimental): Dietary intervention: 210 Kcal, 16g fat, 12g carbohydrate, 2g fibre, 6g sugar, 6g protein
  Interventions: Other: Dietary intervention
- Control 1 (Experimental): Dietary intervention: Water (500 g)
  Interventions: Other: Dietary intervention
- Control 2 (Experimental): Dietary intervention: White bread (190 Kcal, 2g fat, 37g carbohydrate, 2g fibre, 3g sugar, 6g protein)
  Interventions: Other: Dietary intervention
- Control 3 (Experimental): Dietary intervention: Soft baked pretzel (190 Kcal, 2g fat, 38g carbohydrate, 2g fibre, 6g sugar, 4g protein)
  Interventions: Other: Dietary intervention

INTERVENTIONS:
Other: Dietary intervention — All arms are given to all participants, in a randomized order

SUMMARY:
The goal of the proposed research is to investigate the effects of novel snack products differing in macronutrient composition, fibre and sugar content on post-prandial glycemia and short-term appetite control in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking individuals aged 18-55 years with a body mass index of 20.0-29.9 kg/m2

Exclusion Criteria:

* Smokers, individuals with diabetes or other cardiometabolic diseases, persons who suffer from gastrointestinal disorders or have had gastric surgery, or people who regularly use bulk laxatives
* Women with irregular menstruation or who use hormonal contraceptives or hormone replacement therapy
* Individuals who regularly skip breakfast, have allergies to any of the test food ingredients, or who follow a restrictive diet

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-03; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Food intake | 120 minutes
  Food intake (kCal) is assessed 120 min after consumption of the treatments, using an ad libitum pizza lunch design. Participants are asked to eat, during a 20-min period, until feeling comfortably full

SECONDARY OUTCOMES:
Perceived satiety | 120 minutes
  Satiety scores (mm) are assessed using 100-mm "Motivation to Eat" visual analog scale questionnaires. A composite score of the four appetite questions, including Desire to Eat, Hunger, Fullness and Prospective Food Consumption, in the "Motivation to Eat" visual analog scale is calculated to obtain the average appetite score for statistical analysis
Blood glucose | 0 to 120 min (pre-ad libitum lunch) and 140 to 260 min (post-ad libitum lunch) after consumption of treatments
  Blood glucose (mmol/L) is measured using finger prick capillary blood samples
Blood insulin | 0 to 120 min (pre-ad libitum lunch) and 140 to 260 min (post-ad libitum lunch) after consumption of treatments
  Blood insulin (μU/mL) is measured using finger prick capillary blood samples

OTHER OUTCOMES:
Food Recall | 24 hours
  Participants are asked to complete a 24-hour Food Recall starting at dinner the night before each study session and ending at dinner the day of that session.

CONTACTS AND LOCATIONS:
Overall Officials: G. Harvey Anderson, PhD, Principal Investigator — University of Toronto
Locations (1):
- Department of Nutritional Sciences, University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No